CLINICAL TRIAL: NCT01860885
Title: Study of Hospital-wide Critical Respiratory Events Requiring Naloxone in a Pediatric Institution
Brief Title: Critical Respiratory Events in Children Requiring Naloxone: Naloxone Use as Opioid Safety Measure
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN1-2012-1219
Record Dates: First submitted 2013-05-15; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Opioid Induced Respiratory Depression
Keywords: naloxone; children; opioid; respiratory depression; safety
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients requiring naloxone for respiratory depression

SUMMARY:
Opioids are the mainstay of analgesia in hospitalized children but opioid therapy is associated with life-threatening respiratory depression requiring antagonism with naloxone. Hence, it is hypothesized that naloxone requirement can be used as a quality measure of opioid safety. A retrospective medical chart review of 95 patients, who received naloxone for life threatening events, from June 2006-2012, is planned, to identify significant factors associated with risk for opioid induced respiratory depression and formulation of preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* any gender, age or race
* administered naloxone for opioid induced respiratory depression

Exclusion Criteria:

* Any one who did not require naloxone for opioid induced respiratory depression

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who required rescue with naloxone between June 2006 and June 2012; identified based upon an automated trigger report generated from the hospital's risk management database for any dispensation of naloxone from the hospital pharmacy
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Descriptive: Medical history and Risk Factors for critical respiratory events requiring Naloxone in children | about 6 hours around the event
  Data leading to the event and post-event descriptives will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States